CLINICAL TRIAL: NCT03726944
Title: Feasibility of Using a Consumer-based Mobile App to Improve Fatigue and Emotional Symptoms in Myeloproliferative Neoplasm Patients
Brief Title: The Feasibility of Delivering Consumer-based Meditation Applications to Myeloproliferative Neoplasm Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006404
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: This study was a 4-group randomized trial design in which participants were randomly assigned to 4 unique groups that lasted for 8 weeks in total. Each group received two 4-week conditions involving one of three different conditions/arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Meditation1+Meditation2 (Other): 8 weeks in total; 4 weeks of unnamed consumer-based meditation app + 4 weeks of Calm meditation app
  Interventions: Behavioral: Calm App Meditation; Behavioral: Unnamed Consumer-Based App Meditation
- Group 2 - Meditation2+Meditation1 (Other): 8 weeks in total; 4 weeks of Calm meditation app + 4 weeks of unnamed consumer-based meditation app
  Interventions: Behavioral: Calm App Meditation; Behavioral: Unnamed Consumer-Based App Meditation
- Group 3 - Control+Meditation1 (Other): 8 weeks in total; 4 weeks of educational control + 4 weeks of unnamed consumer-based meditation app
  Interventions: Behavioral: Unnamed Consumer-Based App Meditation; Other: Educational Control
- Group 4 - Control+Meditation2 (Other): 8 weeks in total; 4 weeks of educational control + 4 weeks of Calm meditation app
  Interventions: Behavioral: Calm App Meditation; Other: Educational Control

INTERVENTIONS:
Behavioral: Calm App Meditation — The Calm app intervention consisted of 10 min/day of meditation for 4 weeks via the Calm smartphone app.
  Arms: Group 1 - Meditation1+Meditation2; Group 2 - Meditation2+Meditation1; Group 4 - Control+Meditation2
Behavioral: Unnamed Consumer-Based App Meditation — The unnamed consumer-based app intervention consisted of 10 min/day of meditation for 4 weeks via an unnamed consumer-based meditation smartphone app.
  Arms: Group 1 - Meditation1+Meditation2; Group 2 - Meditation2+Meditation1; Group 3 - Control+Meditation1
Other: Educational Control — The educational control consisted of an educational handout that was provided to participants. This control lasted for 4 weeks.
  Arms: Group 3 - Control+Meditation1; Group 4 - Control+Meditation2

SUMMARY:
This study was a four-group randomized pilot trial in myeloproliferative neoplasm (MPN) patients. Patients were recruited nationally through organizational partners and social media. Eligible and consented patients were enrolled into one of four groups, two of which received varying orders of two consumer-based apps (unnamed consumer-based [CB] app and Calm App) and two that received one of the apps alone for the second four weeks of the eight week intervention after an educational control condition. Participants were asked to perform 10 min/day of smartphone-based meditation irrespective of the app and/or the order in which they received the apps. Feasibility outcomes were measured at week five and nine with an online survey. Feasibility outcomes were acceptability, demand, and limited efficacy for depression, anxiety, pain intensity, sleep disturbance, sexual function, quality of life, global health, and total symptom burden. The purpose of this study was to examine the feasibility of the use of two different consumer-based meditation smartphone applications (i.e., apps) in MPN patients.

Specific aim #1: Examine the feasibility of daily meditation delivered using a consumer-based mobile app. Hypothesis: It will feasible to deliver smartphone-based meditation to MPN patients.

Exploratory Aim: Explore the preliminary effects of daily meditation delivered using a consumer-based mobile app on MPN self-report fatigue, anxiety, depression, pain intensity, sleep disturbance, sexual function, global health, quality of life, and total symptom burden. Hypothesis: There will be demonstrated preliminary effects on patient-reported outcomes in MPN patients.

DETAILED DESCRIPTION:
This was a four-group, randomized controlled trial with a cross-over design. Patients were enrolled into one of four groups with varying order of receiving two consumer-based meditation smartphone (i.e., unnamed consumer-based app [CB app], Calm app) apps in 4-week increments over eight weeks. Group #1 received the CB App followed by the Calm app; Group #2 received the Calm app followed by the CB app; Group #3 received educational control followed by the CB app and Group #4 received educational control followed by the Calm app.

MPN patients were recruited online through MPN organizational partners with a single page, broad overview of the study and its requirements. The study was advertised as a smartphone app meditation study. MPN patients interested in the study were asked to complete an online eligibility questionnaire administered via Qualtrics. Researchers then checked completed eligibility questionnaires as they were completed and emailed patients with their eligibility status.

If ineligible, patients received an email stating their ineligibility status as well as links to both consumer-based apps used in the study in case the ineligible participant was interested in trying meditation. Eligible patients were invited to participate in a 20-minute phone appointment in which the study details and informed consent were described in detail. MPN patients who completed the intake appointment were then sent an informed consent electronically via Qualtrics that included a place for their electronic signature.

Upon receipt of the completed informed consent, participants were randomly assigned to one of four groups. A group assignment list was generated prior to study commencement with randomizer.org. This pre-generated list was then used by research personnel to place eligible, consented MPN patients into their group assignment (i.e., Group #1, Group #2, Group #3, Group #4; described below) in the order in which they consented to participate. Randomized participants were provided with a "welcome email" that contained a) a welcome letter introducing them to the study, b) a calendar detailing important study dates, c) instructions specific to the first assigned condition (i.e., CB app, Calm app, or educational control) to be introduced for the first four weeks. After participants completed the first of their two, four-week conditions (i.e., CB App, Calm, or control), they were provided with another email that included instructions specific to their final condition (i.e., CB app, Calm app, or educational control).

Unnamed Consumer-Based (CB) App The CB app was an already existing consumer-based smartphone app. The first and second week consisted of meditation that was basic introductory, and educational for those new to meditation. Weeks three and four consisted of a new and unique daily meditation that study participants could select from a library of meditations within the app. Each of the daily meditations had a different focus (e.g., grief, gratitude, choice, letting go, etc.) and were ~10-12 minutes in length.

Description of Conditions

Calm App The Calm app was an already-existing, consumer-based meditation app. The first week of the intervention included the "7 Days of Calm", which consists of seven days of introductory meditations that incorporated basic, educational information for those new to meditation while introducing brief experiential practices within that short period of time. Weeks two through four consisted of the "Daily Calm", which is a new and unique daily guided meditation that was provided by the app. Each of the daily meditations had a different focus (e.g., practicing patience, loving-kindness, gratitude, etc.) and were ~10-12 minutes in length.

Educational Control The control condition was provided with educational material handout that was developed by the research team prior to the study. The handout addressed MPN patient fatigue (e.g., What causes fatigue?) as well as examples of and information related to evidence-based fatigue-management strategies.

Description of Groups

Group #1 (CB App + Calm) Group #1 was assigned the CB App (Weeks 1-4) and the Calm app (Weeks 5-8). During weeks 1-4, participants were asked to complete four weeks of meditation on the CB App via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could. During weeks 5-8, participants were asked to complete four weeks of meditation on the Calm app via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could.

Group #2 (Calm APP + CB App) Group #2 was assigned the Calm app (Weeks 1-4) and the CB app (Weeks 5-8). During weeks 1-4, participants were asked to complete four weeks of meditation on the Calm app via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could. During weeks 5-8, participants were asked to complete four weeks of meditation on the CB app via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could.

Group #3 (Control + CB App) Group #3 was assigned educational control (Weeks 1-4) and the CB app (Weeks 5-8). During weeks 1-4, participants were provided the educational material handout and asked to maintain their normal routine. During weeks 5-8, participants were asked to complete four weeks of meditation on the CB app via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could.

Group #4 (Control + Calm) Group #4 was assigned educational control (Weeks 1-4) and the Calm app (Weeks 5-8). During weeks 1-4, participants were provided the educational material handout and asked to maintain their normal routine. During weeks 5-8, participants were asked to complete four weeks of meditation on the Calm app via their smartphone for a minimum of 10 min/day (i.e., ~70 min/week) but encouraged to do more if they could.

All study participants completed patient-reported outcomes measures via an online questionnaire at baseline (week 0), mid-point (week 5), and post-intervention (week 9).

ELIGIBILITY:
Inclusion Criteria:

* had a diagnosis of MPN (i.e., essential thrombocythemia, polycythemia vera, or myelofibrosis) identified by treating physician
* owned a mobile smartphone and were willing to download and use a meditation app (i.e., CB or Calm)
* could read and understand English
* were age 18 years or older
* were willing to be randomized to one of four groups: 1) CB 4 wks/Calm 4 wks, 2) Calm 4 wks/CB 4 wks, 3) educational material 4 wks/CB 4 wks, and 4) educational material 4 wks/Calm 4 wks,

Exclusion Criteria:

* engaged in ≥10 min/day of meditation on ≥5 days/week for the past 6 months
* engaged in ≥60 min/week of tai chi, qigong, or yoga each week
* utilized either App #1 or Calm
* resided outside of the United States of America

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention: survey | Change from Baseline to Week 5 and Week 9
  Acceptability was measured with a satisfaction survey. Benchmarks for acceptability included ≥70% response to the following questions in the survey: 1) satisfaction with the apps' content, 2) intending to continue using the app, 3) enjoying using the apps, and 4) recommending it for other MPN patients. The % of participants indicating responses to the four prior questions will be considered "acceptable" if all four questions are responded to with a ≥70% response rate.
Demand of Meditation | Change from Baseline to Week 5 and Week 9
  Demand was measured using adherence to the meditation intervention. Meditation participation was tracked by the smartphone app developers and reported to the Principal Investigator. Adherence benchmarks were defined as an average of ≥49 min/week of meditation across all participants (i.e., ≥70% of prescribed meditation).
Limited-Efficacy Testing of Meditation | Change from Baseline to Week 5 and Week 9
  Limited-efficacy testing was measured with Cohen's d effect sizes calculated for patient-reported outcomes (described below as secondary outcomes).

SECONDARY OUTCOMES:
MPN Total Symptom Burden (severity and symptomology) | Change from Baseline to Week 5 and Week 9
  A 10-item, validated form that calculates total symptom burden score (MPN Symptom Assessment Form Total Symptom Score). A higher score indicates a worse MPN-specific symptom burden; scores range from 0-100
Fatigue | Change from Baseline to Week 5 and Change from Baseline to Week 9
  A single-item fatigue question taken from the MPN Symptom Assessment Form; scores can range from 0-10
Anxiety | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Anxiety Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 36.3-82.7
Depression | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Depression Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 41.0-79.4
Sleep Disturbance | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Sleep Disturbance Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 32.0-73.3
Sexual Function | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Sexual Function consisting of five sub-scales; these scales consist of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; the five sub-scales include vaginal discomfort (score range of 33.2-77.08), lubrication (score range of 30.99-69.26), erectile function (score range of 30.72-68.47), satisfaction with sex life (score range of 29.59-72.01), and interest in sexual activity (score range of 32.02-76.17)
Pain Intensity | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Pain Intensity Adult Short Form; this scale consists of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; scores range from 30.7-71.8
Global Health | Change from Baseline to Week 5 and Week 9
  National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Global Health consisting of Physical Health and Mental Health sub-scales; these scales consist of a series of questions that are tallied up into a sum score and converted to a standardized t-score. A higher score represents a higher presence, not necessarily a better or worse score, of the item being measured; score ranges for physical health are 16.2-67.7 and score ranges for mental health are 21.1-67.6

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Huberty J, Eckert R, Larkey L, Kurka J, Rodriguez De Jesus SA, Yoo W, Mesa R. Smartphone-Based Meditation for Myeloproliferative Neoplasm Patients: Feasibility Study to Inform Future Trials. JMIR Form Res. 2019 Apr 29;3(2):e12662. doi: 10.2196/12662. PMID 31033443